CLINICAL TRIAL: NCT01360801
Title: High Definition White Light Endoscopy and Narrow Band Imaging for the Assessment of Barrett's Disease After Endoscopic Therapy
Status: Terminated | Type: Observational
Why Stopped: enrollment moved very slowly which was not anticipated, and, funding issues
Sponsor: Mayo Clinic (Other)
Collaborators: Olympus (Industry)
Responsible Party: Principal Investigator, Herbert C. Wolfsen, Professor of Medicine, Mayo College of Medicine; Director of Endoscopy, Mayo Clinic Florida, Mayo Clinic
Other Study IDs: 10-003234
Record Dates: First submitted 2011-05-18; First posted 2011-05-26 (Estimated); Last update posted 2014-04-10 (Estimated); Status verified 2014-04

CONDITIONS: Barrett's Esophagus
MeSH Terms: conditions — Barrett Esophagus

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The investigators seek to test the hypothesis that the improved version of high definition white light endoscopes and Narrow Band Imaging (NBI) are more accurate in detecting residual Barrett's Metaplasia and Dysplasia disease after previous resection or ablation treatments than current versions of these endoscopes.

DETAILED DESCRIPTION:
Information will be collected. Images will be taken.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years and older
* Patients with Barrett's esophagus (BE) dysplasia as the original indication for treatment
* Undergoing any type of endoscopic BE resection or ablation treatment including RFA, cryotherapy, photodynamic therapy, or EMR, or combinations of these.
* <1cm of circumferential, peninsular, or island-type BE on prior endoscopy or ablation
* Ability to provide written, informed consent

Deferral Criteria: This category is for patients in two specific situations, 1) Erosive esophagitis, and, 2) presence of a nodule suspicious for the presence of neoplasia.

1. Erosive esophagitis: patients found to have erosive esophagitis, will be deferred for up to 3 months from their Index study procedure, to permit more aggressive medical therapy to heal the erosive esophagitis. After healing, the Index study procedure will be performed up to 3 months later, and the follow-up endoscopy (and study closure) performed 3 to 6 months after that (total of no more than 9 months).
2. Presence of nodule suspicious for neoplasia: for patients found to have such nodular lesions, the Index study procedure will be deferred for 3 months, while Endoscopic Mucosal Resection is performed and subsequently heals.

Note: Only one deferral per patient is permitted, and this one deferral is allowed only for these specific criteria. The end of the study will be defined by the time of follow-up of the last patient who was not deferred; any deferred patients who have not completed follow-up procedures by that time, may miss their follow-up visit as part of the study. (This is to prevent the possibility of delaying the close of the study due to deferral of a procedure late in the study.)

Exclusion Criteria:

* Current participation in another clinical study
* Complete eradication of BE documented by biopsies in 3 or more previous endoscopic procedures performed after resection/ablation
* Inability to obtain biopsies due to anticoagulation, varices, etc.
* Pregnancy
* Worse than Grade C erosive esophagitis
* Less than 3 weeks from previous endoscopy with biopsy or 6 weeks from previous endoscopic therapy (ablation or resection).

Ages: 18 Years to 88 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Men and women (not pregnant) presenting to the GI Lab for Upper Endoscopy. Child-bearing potential not excluded.
Sampling Method: Non-Probability Sample
Enrollment: 21 (Actual)
Dates: Start 2011-02; Primary Completion 2014-03 (Actual); Study Completion 2014-03 (Actual)

PRIMARY OUTCOMES:
Accuracy of Agreement Between Imaging and Histology | 9 months
  The accuracy of agreement between endoscopic imaging diagnosis compared with biopsy histology diagnosis.

SECONDARY OUTCOMES:
Presence of Residual Disease | 9 months
  Presence of any residual Barrett's disease at follow-up endoscopy after ablation / resection treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Herbert C. Wolfsen,, M.D., Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic, Jacksonville, Florida, United States